CLINICAL TRIAL: NCT00001891
Title: Assessment of Myocardial Viability Utilizing Myocardial Contrast Echocardiography
Brief Title: Myocardial Contrast Echocardiography (MCE) to Check for Living and Working Heart Muscle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990108; 99-H-0108
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-03

CONDITIONS: Coronary Disease; Heart Diseases
Keywords: CABG; Hibernation; LV Function; Microbubbles; Revascularization; Coronary Artery Disease
MeSH Terms: conditions — Coronary Disease; Heart Diseases; Coronary Artery Disease

INTERVENTIONS:
Procedure: Myocardial contrast echocardiography
Procedure: Dobutamine echocardiography

SUMMARY:
Coronary artery disease (CAD) can cause poor blood flow and supply to the heart muscle. It can result in irreversible damage to the heart muscle and poor function. Before treating patients with heart disease it is important to know how well the heart is functioning. Echocardiography is a diagnostic test that can measure heart function. If part of the heart muscle is not working properly due to previous damage, echocardiography can provide information about how much improvement can be expected after treatment (surgery or angioplasty).

The purpose of this study is to compare the accuracy of myocardial contrast echocardiography (MCE) to dobutamine echocardiography to detect the potential for damaged heart muscle to be treated and function in patients with heart disease.

Myocardial contrast echocardiography (MCE) does not use radioactivity. It uses sound waves like standard echocardiography. However, with MCE patients receive an injection of a "contrast agent" directly into the blood stream through a vein. The contrast agent, called Optison, is made of tiny microbubbles smaller than red blood cells. The echocardiogram can detect these microbubbles in the small blood vessels of the heart muscle and allow researchers to find areas of the heart receiving less blood flow than others.

Echocardiography with Dobutamine does not use radioactivity. It uses sound waves, like standard echocardiography. During this echocardiogram patients receive doses of a medication called dobutamine that stimulates the heart to beat stronger and faster. Heart muscle that does not beat stronger after dobutamine is probably dead, usually as a result of a previous heart attack.

DETAILED DESCRIPTION:
Dobutamine echocardiography has become a valuable technique for the evaluation of myocardial viability in patients with coronary artery disease (CAD) and dysfunctional myocardium because it can accurately predict which myocardial segments will show contractile recovery after successful revascularization. Myocardial contrast echocardiography (MCE) offers the potential to evaluate tissue perfusion at the level where oxygen transfer to the myocytes occurs. MCE, therefore, can provide information regarding the functional status of the myocardial microvasculature which has a close relationship with myocellular integrity. The purpose of this study is to evaluate the accuracy of MCE compared to dobutamine echocardiography to detect myocardial viability in patients with CAD and resting wall motion abnormalities.

ELIGIBILITY:
Patients undergoing evaluation for CAD who show at least two myocardial segments with wall motion abnormalities on a baseline echocardiogram will be offered to participate in this study.

Patients will be adults older than 21 years of age.

No pre-menopausal patients who are lactating, are pregnant or potentially pregnant as judged by history, physical examination, ultrasound or urine pregnancy test.

No one with unstable angina.

No subjects with recent myocardial infarction (less than 1 month).

No one with frequent ectopy which precludes adequate imaging acquisition.

No subjects with significant hypertension (systolic blood pressure greater than 170 mm Hg).

No hypotension with basal sitting systolic arterial pressure less than 100 mm HG confirmed 30 minutes later.

No subjects with sinus tachycardia greater than or equal to 100 beats/minute.

No atrial fibrillation.

No inadequate two-dimensional echocardiographic windows.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1999-05; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Maisey M. Evaluating the benefits of nuclear cardiology. Q J Nucl Med. 1996 Mar;40(1):47-54. PMID 8681013
- [Background] Vanoverschelde JL, Wijns W, Depre C, Essamri B, Heyndrickx GR, Borgers M, Bol A, Melin JA. Mechanisms of chronic regional postischemic dysfunction in humans. New insights from the study of noninfarcted collateral-dependent myocardium. Circulation. 1993 May;87(5):1513-23. doi: 10.1161/01.cir.87.5.1513. PMID 8491006